CLINICAL TRIAL: NCT02721290
Title: Comparison of the Sensitive Cutaneous Block Distribution Following Femoral Nerve Block Using an Ultrasound Plus Neurostimulator Technique Versus an Approach Based on the Localization of the Femoral Artery.
Brief Title: Comparison of the Sensitive Cutaneous Block Distribution Following Femoral Nerve Block Using Two Femoral Block Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Issam TANOUBI, Associate professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160112
Record Dates: First submitted 2016-03-15; First posted 2016-03-29 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Regional Anesthesia; Femoral Nerve Block
Keywords: Knee surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block using Ultrasound and neurostimulator (Active Comparator): Femoral block using the standard technique of ultrasound for femoral nerve identification and neurostimulator set at between 0.3-0.5 mA with quads muscle response for needle placement confirmation before injecting 20cc of Ropivacaine 0.5%.
  Interventions: Procedure: Femoral nerve block using Ultrasound and neurostimulator; Drug: Ropivacaine 0.5%
- Femoral nerve block using femoral artery target (Experimental): Femoral block using the alternate technique of aiming for the inferolateral aspect of the femoral artery and injecting 20cc of Ropivacaine 0.5%.
  Interventions: Procedure: Femoral nerve block using Ultrasound; Drug: Ropivacaine 0.5%

INTERVENTIONS:
Procedure: Femoral nerve block using Ultrasound and neurostimulator
  Arms: Femoral nerve block using Ultrasound and neurostimulator
Procedure: Femoral nerve block using Ultrasound
  Arms: Femoral nerve block using femoral artery target
Drug: Ropivacaine 0.5% — Ropivacaine 0.5% (20cc total) will be injected for the performance of the block in the two arms of the study.

SUMMARY:
In this study, we will be comparing two approaches to the femoral block. The first or classical approach and one that is the most popular in our institution is used by combining ultrasound guidance and neurostimulator to do the block. The second is performed with the ultrasound alone aiming at the inferolateral aspect of the femoral artery with the needle and injecting. The primary endpoint of the study is the sensitive cutaneous block distribution using both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an elective surgery for which the anesthesiologist planned to do a single shot or continuous femoral nerve block.

Exclusion Criteria:

* Any contraindication to the femoral nerve block (coagulopathy, infection, pre-existing neuropathy, local anesthetic allergy and refusal of local anesthesia).
* Refusal to participate in the study
* Inability to understand or communicate the effect of local anesthesia secondary to the femoral nerve bloc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sensitive cutaneous block distribution area for the two techniques | 45 minutes
  After performance of a femoral nerve block, ice will be applied on the skin to plot the anesthetized area at times 15, 30 and 45 mn. The sensation will be compared on a scale from 0 (no sensation) to 2 (no anesthesia) with the contralateral leg. An area in cm2 will be calculated for each of the patients and the two techniques will then be compared.

SECONDARY OUTCOMES:
Time of block completion | 45 minutes
  Time recorded from the end of the cutaneous local anesthetic injection to the end of the 20cc injection of the 0.5% Ropivacaine (time of block completion)
Ease of ultrasound visualization of the femoral nerve | 45 minutes
  This will be assessed by the anesthesiologist making the femoral nerve block from a scale of 1 (no visualization) to 10 (excellent visualization).
Ease of ultrasound visualization of the femoral artery | 45 minutes
  This will be assessed by the anesthesiologist making the femoral nerve block from a scale of 1 (no visualization) to 10 (excellent visualization).
Numbers of needle redirection | 45 minutes
  The number of time for each patients using either techniques that the needle will have been withdrawn.
Vascular puncture | 45 minutes
  Presence or absence of blood return at anytime in the tubing while performing the block.
Paresthesia | 45 minutes
  Presence or absence of the sensation of electrical shock felt by the patient in the territory of the femoral nerve at any point while performing the block
Patient Satisfaction | 45 minutes
  Satisfaction expressed by the patient after the completion of the femoral nerve block using a scale from 1 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada